CLINICAL TRIAL: NCT03212248
Title: CRP (C-Reactive-Protein) and Pneumonia Biomarkers Stratification for Selectively Addressing Priorities in Thoracic Emergency Ultrasound in Pneumonia
Brief Title: CRP and Thoracic Emergency Ultrasound in Pneumonia
Acronym: TUS-STRAT
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Collaborators: Ospedale Civile di Ragusa, Italy (Unknown)
Responsible Party: Principal Investigator, Guglielmo Trovato, MD, PhD, Professor of Medicine - Research Project Planning Unit, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Other Study IDs: TUS-STRAT
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Difference, Individual; Community-acquired Pneumonia; Ultrasound
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thoracic Ultrasound (TUS)

SUMMARY:
This preliminary study investigates in patients with possible clinical diagnosis of pneumonia, clues and biomarker assessed at Emergency Department (ED) triage, potentially predicting detection of lung consolidation by Thoracic-ultrasound (TUS) and/or by Chest-X-Rays. Cough and high admission CRP levels will be defined according to the cutoff defined by ROC analysis, will be challenged if independently associated with TUS lung consolidation detection High level of the chosen biomarker, and any of the considered symptoms, in otherwise not extremely critical patients (CURB65≤3), should prompt to immediate confirm by TUS, during the physical examination. This may limit the need of further radiological investigations allowing targeted workup.

DETAILED DESCRIPTION:
Chest-X-Rays (CXR), Computerized Tomography (CT) or Thoracic Ultrasound (TUS) provide images deemed consistent with acute lung consolidation and suitable to confirm the diagnosis of community acquired pneumonia (CAP). Patients which may be affected by CAP are many , but diagnosis is not straightforward because we are managing "a disease characterized by educated guesswork" . Comprehensive imaging workup may be not regularly affordable in busy emergency rooms. Point-of-care TUS allows reliable diagnosis of lung consolidation and of pleural effusion. Regretfully, adequate TUS expertise is more warranted than actually available in most medical departments. Even not specifically investigated, a delay or even an impairment of appropriate TUS or CXR evaluation for several patients may occur due to time- or resource-limiting factors.

Clinical clues of lung consolidation are many. Key symptoms are cough, fever, chest pain and dyspnea with tachypnea, while the major physical signs are chest crackles and dullness. Surrogate biomarkers more easily obtainable in emergency facilities are C-reactive-protein (CRP), peripheral non-invasive pulse-oxymetry and neutrophil-to-lymphocyte ratio (NLR) which is an index of systemic inflammation associated also with pneumonia and subsequent outcome.

The aim of this preliminary study is to evaluate if any clue and which biomarker, including NLR, assessed at Emergency Department (ED) triage, is predictive of the subsequent detection of lung consolidation by TUS and/or by CXR.

The minimal groups' size, with and without TUS or CXR lung consolidation, was calculated according to the difference of the averages of neutrophil-to-lymphocyte ratio (NLR) in the reference the study of Yoon et al. Accepting alpha 0.01, for the probability of type 1 error, and power 80% for probability of type 2 error, a minimum sample size of 19 participants in each group (total 38) was required. Student's t-tests assessed the differences of CRP, WBC - white blood cells count - (TLC), neutrophil count (TNC) and NLR, between the groups with TUS and, separately, with CXR lung consolidation.Thereafter, by ROC (receiver operating curve) analysis, a cutoff of NLR, total leucocytes count (TLC), total Neutrophil count (TNC) and of CRP was calculated vs. the optimal reliability for the detection of TUS consolidation; sensitivity, specificity and accuracy (The proportion of all tests that are correct), and relative Odds Ratio (OR) and confidence intervals (CI) of the individual symptoms, and ORs of so defined laboratory assay cut-offs were calculated separately vs. TUS and CXR consolidation.

ELIGIBILITY:
Inclusion Criteria:

presence of history and symptoms, signs at physical examination and early laboratory clues of CAP According to the preliminary triage, in all patients, as a routine assessment, breath frequency, blood pressure and heart rate, pulse oxymetry, serum and blood analysis including creatinine and urea, CRP, blood cell counts and hemoglobin assay, were performed, also for CURB65 staging. ECG was preliminary done in all patients with chest pain, dyspnea and/or fever.

Exclusion Criteria:

-

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criteria of exclusion: severe respiratory failure - pulse oxymetry ≥92%, myocardial infarction, acute pulmonary edema or severe heart failure, excluded on clinical basis, severe COPD excluded by patient's history and by subsequent CXR, CURB65 ≥3.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Odds of detecting lung consolidation by TUS according to symptoms or biomarkers' cutoffs | ten minutes
  ultrasound

SECONDARY OUTCOMES:
Odds of detecting lung consolidation by Chest X Rays (CXR) according to symptoms or biomarkers' cutoffs | ten minutes
  radiology

CONTACTS AND LOCATIONS:
Overall Officials: GUGLIELMO TROVATO, MD, Study Chair — medint
Locations (1):
- MCAU, Catania, Please Select An Option Below, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Interrigi MC, Trovato FM, Catalano D, Trovato GM. Emergency thoracic ultrasound and clinical risk management. Ther Clin Risk Manag. 2017 Feb 9;13:151-160. doi: 10.2147/TCRM.S126770. eCollection 2017. PMID 28223817
- [Background] Sperandeo M, Rea G, Grimaldi MA, Trovato F, Dimitri LM, Carnevale V. Contrast-enhanced ultrasound does not discriminate between community acquired pneumonia and lung cancer. Thorax. 2017 Feb;72(2):178-180. doi: 10.1136/thoraxjnl-2016-208913. Epub 2016 Oct 14. PMID 27742872
- [Background] Trovato FM, Catalano D, Trovato GM. Thoracic ultrasound: An adjunctive and valuable imaging tool in emergency, resource-limited settings and for a sustainable monitoring of patients. World J Radiol. 2016 Sep 28;8(9):775-784. doi: 10.4329/wjr.v8.i9.775. PMID 27721940
- [Background] Trovato FM, Catalano D. Diagnosis of Pneumonia by Lung Ultrasound in Children and Limited Resources Subsets: A Valuable Medical Breakthrough. Chest. 2016 Jul;150(1):258-60. doi: 10.1016/j.chest.2016.04.032. No abstract available. PMID 27396790
- [Background] Waterer GW. The Diagnosis of Community-acquired Pneumonia. Do We Need to Take a Big Step Backward? Am J Respir Crit Care Med. 2015 Oct 15;192(8):912-3. doi: 10.1164/rccm.201507-1460ED. No abstract available. PMID 26469839
- [Background] Cataudella E, Giraffa CM, Di Marca S, Pulvirenti A, Alaimo S, Pisano M, Terranova V, Corriere T, Ronsisvalle ML, Di Quattro R, Stancanelli B, Giordano M, Vancheri C, Malatino L. Neutrophil-To-Lymphocyte Ratio: An Emerging Marker Predicting Prognosis in Elderly Adults with Community-Acquired Pneumonia. J Am Geriatr Soc. 2017 Aug;65(8):1796-1801. doi: 10.1111/jgs.14894. Epub 2017 Apr 13. PMID 28407209
- [Background] Yoon NB, Son C, Um SJ. Role of the neutrophil-lymphocyte count ratio in the differential diagnosis between pulmonary tuberculosis and bacterial community-acquired pneumonia. Ann Lab Med. 2013 Mar;33(2):105-10. doi: 10.3343/alm.2013.33.2.105. Epub 2013 Feb 21. PMID 23482854